CLINICAL TRIAL: NCT04826159
Title: A Pharmacodynamic Study to Evaluate the Effects of IMB-1018972 on Myocardial Energetics, Metabolism, and Function in Patients With Type 2 Diabetes.
Brief Title: IMPROVE-DiCE: Study to Evaluate Effect of IMB-1018972 on Cardiac Energetics in T2DM & Obesity (Pt 1) With HFpEF (Pt 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imbria Pharmaceuticals, Inc. (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMB101-005
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; Diabetic Cardiomyopathies; HFpEF - Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IMB-1018972 200 mg (Experimental)
  Interventions: Drug: IMB-1018972

INTERVENTIONS:
Drug: IMB-1018972 — Modified release tablet for oral administration

SUMMARY:
The purpose of this study is to assess the activity of IMB-1018972 on cardiac energetic reserve at rest and during stress and to assess safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Elevated HbA1c
* Elevated BMI
* Preserved left ventricular ejection fraction
* Diagnosis of HFpEF (Stage 2 only)

Exclusion Criteria:

* Uncontrolled hypertension
* Contraindication to magnetic resonance scanning
* More than mild to moderate valvular heart disease
* Atrial fibrillation
* History of sustained ventricular tachycardia or cardiac arrest
* Inability to exercise (Stage 2 only)
* Clinically significant concurrent condition which could prevent the patient from performing any of the protocol-specified assessments, represent a safety concern if the patient participates in the trial or could confound trial assessments of safety or tolerability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Change in cardiac PCr/ATP ratio at rest (Stage 1 and Stage 2) measured by 31P-MRS at baseline and at EOT with 200 mg BID of IMB-1018972. | Baseline, End of Treatment (up to 16 weeks)
Change in cardiac PCr/ATP ratio with dobutamine stress (Stage 1 only) measured by 31P-MRS at baseline and at EOT with 200 mg BID of IMB-1018972 | Baseline, End of Treatment (up to 8 weeks)

SECONDARY OUTCOMES:
Safety and tolerability of IMB-1018972 as measured by incidence and severity of treatment emergent AEs (including AEs leading to study drug discontinuation and AEs leading to death), as well as incidence of treatment emergent SAEs | Baseline through End of Treatment (up to 16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Yavari, BSc, MBBS, DPhil, Study Chair — Imbria Pharmaceuticals, Inc.
Locations (1):
- Oxford University Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hundertmark MJ, Birkhoelzer SM, Portwood C, Siu AG, Matthews V, Lewis AJ, Grist J, Mozes F, Henry JA, Patel J, Chamberlin P, Sarwar R, Yavari A, Dehbi HM, Rao P, Shi X, Zheng S, Robbins JM, Gerszten RE, Frenneaux MP, Valkovic L, Miller JJJJ, Neubauer S, Tyler DJ, Rider OJ. IMPROVE-DiCE, a 2-Part, Open-Label, Phase 2a Trial Evaluating the Safety and Effectiveness of Ninerafaxstat in Patients With Cardiometabolic Syndromes. Circulation. 2025 Dec 18. doi: 10.1161/CIRCULATIONAHA.125.074041. Online ahead of print. PMID 41410037